CLINICAL TRIAL: NCT06170710
Title: Postoperative Concurrent Chemoradiotherapy Followed by Anti-PD-1 Antibody Maintenance Therapy in High-Risk Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Postoperative CCRT Followed by Immunotherapy in High-Risk LA HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23/219-3961
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT+ cisplatin+Anti-PD-1 antibody (Experimental): Concurrent cisplatin-RT followed by PD-1 antibody
  Interventions: Drug: Anti-PD-1 monoclonal antibody; Other: Postoperative CCRT
- RT+ cisplatin (Active Comparator): Concurrent cisplatin-RT
  Interventions: Other: Postoperative CCRT

INTERVENTIONS:
Drug: Anti-PD-1 monoclonal antibody — Postoperative CCRT followed by any anti-PD-1 monoclonal antibody of the following:
  Pembrolizumab, 200mg, Q3W or Nivolumab, 3mg/kg, Q2W or Tislelizumab，200mg，Q3W or Camrelizumab，200mg，Q3W or Sintilimab，200mg，Q3W or Toripalimab，240mg，Q3W
  Arms: RT+ cisplatin+Anti-PD-1 antibody
Other: Postoperative CCRT — Postoperative chemoradiotherapy

SUMMARY:
This trial aims to evaluate whether the addition of anti-PD-1 antibody to adjuvant postoperative chemoradiotherapy could improve disease free survival in patients with high-risk locally advanced head and neck squamous cell carcinoma (HNSCC).

DETAILED DESCRIPTION:
This open-label, randomized, controlled, phase II study will include 173 patients who have been operated for their LA SCCHN with high risk.

Subjects will be randomized (1:1) to receive post-operative concomitant cisplatin-RT followed by/not PD-1 antibody.

The study is designed with the general objective of demonstrating that treatment CCRT followed by PD-1 antibody is more efficient than CCRT alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the head and neck which include but not limit following primary sites: oral cavity, oropharynx, hypopharynx or larynx
* Patients eligible with one or more High-Risk factors of the following: For HPV+ OPSCC: T4 OR cN3 OR pN2 OR non-R0 resection OR resection margin<5mm OR ENE (+) OR perineural invasion OR vessel/lymphatic vessel invasion；For HPV- HNSCC：T4 OR cN3 OR pN2 OR non-R0 resection OR resection margin<5mm OR ENE (+) OR perineural invasion OR vessel/lymphatic vessel invasion OR IV/V cervical lymph node metastases
* ECOG performance score 0-1
* PD-L1 expression with CPS>1
* No contraindications to immunotherapy or chemoradiotherapy
* Adequate organ function
* Female subject of childbearing potential should have a negative pregnancy test within 7 days prior to receiving the first dose of study medication.Female subjects of childbearing potential must be willing to use an adequate method of contraception during the course of the study and 60 days after the last dose of study medication.
* Reproductive male subjects must agree to use an adequate method of contraception during the course of the study and 60 days after the last dose of study medication.
* Informed consent is obtainable.

Exclusion Criteria:

* Previous or co-existing malignancies, except cured basal cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer
* Active infection
* Known active viral infection Human Immunodeficiency Virus (HIV), Hepatitis B/C) or known history of positive test for HIV
* Active and/or historical autoimmune disease, except patients with vitiligo or asthma that has completely resolved in childhood and does not require any intervention in adulthood
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
* Pregnant, breastfeeding patients, and female patients of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception as outlined in the protocol for the duration of the study
* History of PD-1/L1 treatment
* If the subjects underwent major surgery for non-tumors, the toxicity and complications of the surgery needed to be adequately treated and the body conditions returned to normal
* Concurrent enrollment in another clinical trial using an investigational anti-cancer treatment within 28 days prior to the first dose of study treatment
* Other circumstances leading to the termination of the study, as determined by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Disease free survival at year 2 (2y-DFS) | From randomization until time of events up to 2 years
  Disease-free survival time is defined as the time from date of randomization until the first disease recurrence（including carcinoma in situ）or death from any cause.

SECONDARY OUTCOMES:
Locoregional control at year 2 (2y-LRC) | From randomization until time of events up to 2 years
  LRC defined from randomization to first radiographically or pathologically confirmed local or regional recurrence.
Overall survival at year 2 (2y-OS) | From randomization until death due to any cause, up to 2 years
  Time between the date of randomization and death.
Adverse events | From randomization until time of events up to 2 years
  Adverse events and serious adverse events according to CACTE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jingbo Wang, Dr., Principal Investigator — National Cancer Cencer/Cancer hospital
Locations (1):
- National Cancer Cencer/Cancer hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No